CLINICAL TRIAL: NCT00416117
Title: The Effectiveness of Manual Physical Therapy and Exercise for Mechanical Neck Disorders: A Randomized Controlled Trial
Brief Title: Manual Physical Therapy and Exercise for Mechanical Neck Disorders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: 59th Medical Wing (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.2001.123
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2006-12-27 (Estimated); Status verified 2006-12

CONDITIONS: Neck Pain; Radiculitis
Keywords: Neck pain; Cervical pain; Radicular pain; Manual therapy; Mobilization; Manipulation
MeSH Terms: conditions — Neck Pain; Radiculopathy | interventions — Exercise

INTERVENTIONS:
Procedure: Manual Physical Therapy and Exercise
Procedure: Minimal Intervention

SUMMARY:
Mounting evidence does support the combined use of manual physical therapy (MPT)and exercise for patients with cervicogenic headache and mechanical neck pain. However, there is insufficient evidence to assess the effectiveness of MPT and exercise for patients with neck disorders with radicular symptoms. Our purpose for this study was to determine the effectiveness of a manual physical therapy and exercise program as compared to a minimal intervention approach in the treatment of patients with mechanical neck pain, with or without upper extremity symptoms.

DETAILED DESCRIPTION:
Prior to randomization, potential participants underwent a standardized history and examination of the cervical spine and upper quarter. We collected demographic information that included each patient's age; gender; medication use; imaging results; and the location, nature, and duration of symptoms. Self-report measures included the NDI and VAS pain scales. Physical exam measures included cervical range of motion measurements with a gravity inclinometer, passive accessory motion testing to assess cervical spine segmental mobility and pain provocation, an upper quarter neurological screening, and special tests commonly used to identify cervical impairments.

Participants meeting all inclusion criteria were randomized into one of two treatment groups: 1) manual physical therapy and exercise (MTE) or 2) minimal intervention (MI).

Patients in the MTE group received manual physical therapy interventions specifically targeted to impairments identified during the physical examination. Physical therapists chose manual interventions consisting of thrust and non-thrust joint manipulation/mobilization, muscle energy, and soft-tissue mobilization/stretching techniques that are commonly referenced and used in clinical practice. We provided all patients in the MTE group with a standard home exercise program of cervical retraction, deep neck flexor strengthening, and cervical rotation range of motion exercises.

Patients in the MI group received a basic treatment plan consistent with general practitioner care. We provided all patients with a basic regimen of postural advice, encouragement to maintain neck motion and daily activity levels, cervical rotation range of motion exercise, and instructions to continue any prescribed medication use. Minimalist physical therapy treatments consisted of sub-therapeutic pulsed (10%) ultrasound at 0.1w/cm2 for 10 minutes applied to the cervical spine and cervical rotation range of motion exercises. We provided these treatments to maintain the patients' expectations for physical therapy treatment and subsequent improvement, and to standardize the therapist-patient interaction time

The intervention period lasted 3 weeks with both groups receiving treatment twice weekly for up to 6 sessions. We standardized treatment time for both groups by using a one-hour initial evaluation and treatment session and thirty-minute follow-up treatment sessions. Patients did not have to complete all six visits if their symptoms had fully resolved. The treating therapist instructed and supervised all exercises to ensure proper patient technique and understanding.

We collected outcome measure data at baseline and at the patient's 3-week, 6-week and 1-year follow-ups. All outcome measures were collected by physical therapists that were blinded to treatment group allocation.

ELIGIBILITY:
Inclusion Criteria:

* primary complaint of neck pain, with or without unilateral upper extremity symptoms
* age greater than 18
* Neck Disability Index (NDI) score greater than or equal to 10 points
* Composite Visual Analog Scale (VAS) score greater than or equal to 30mm
* Eligible for military health care
* Reside within one hour of the military treatment facilities
* Possess sufficient English language skills to complete all questionnaires

Exclusion Criteria:

* whiplash injury within the past 6 weeks
* history of spinal tumors, spinal infection, cervical spine fracture, or previous neck surgery
* pending legal action regarding their neck pain
* diagnosis of central cervical spinal stenosis
* bilateral upper extremity symptoms
* two positive neurological findings at the same nerve root level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-07; Study Completion 2004-06

PRIMARY OUTCOMES:
Neck Disability Index
Visual analog scale for neck pain
Visual analog scale for upper extremity pain
Global rating of change

SECONDARY OUTCOMES:
Treatment success rates based on GRC
Additional healthcare utilization

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Walker, PT, DSc, Principal Investigator — Brooke Army Medical Center
Locations (2):
- United States (2):
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas

REFERENCES:
- [Derived] Walker MJ, Boyles RE, Young BA, Strunce JB, Garber MB, Whitman JM, Deyle G, Wainner RS. The effectiveness of manual physical therapy and exercise for mechanical neck pain: a randomized clinical trial. Spine (Phila Pa 1976). 2008 Oct 15;33(22):2371-8. doi: 10.1097/BRS.0b013e318183391e. PMID 18923311